CLINICAL TRIAL: NCT01877889
Title: A Double-Blind, Randomized, 2-Way Crossover Study to Compare the Pharmacodynamics of Canagliflozin 300 mg Versus Dapagliflozin 10 mg in Healthy Subjects
Brief Title: A Study to Compare the Pharmacodynamics of Canagliflozin and Dapagliflozin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR101974; 28431754DIA1056 (Other: Janssen-Cilag International NV); 2013-000994-54 (EudraCT Number)
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin; INVOKANA; Dapagliflozin; FORXIGA; Pharmacodynamics
MeSH Terms: interventions — Canagliflozin; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: Cana (Experimental): Each volunteer will receive 300 mg of canagliflozin once daily for 4 days.
  Interventions: Drug: Canagliflozin
- Part 2: Sequence 1 (Dapa/Cana) (Experimental): Each volunteer will receive 10 mg of dapagliflozin once daily for 4 days (treatment period 1) followed by 300 mg of canagliflozin once daily for 4 days (treatment period 2). Each treatment period will be separated by a 12- to 14-day washout period (with no medication).
  Interventions: Drug: Canagliflozin; Drug: Dapagliflozin
- Part 2: Sequence 2 (Cana/Dapa) (Experimental): Each volunteer will receive 300 mg of canagliflozin once daily for 4 days (treatment period 1) followed by 10 mg of dapagliflozin once daily for 4 days (treatment period 2). Each treatment period will be separated by a 12- to 14-day washout period.
  Interventions: Drug: Canagliflozin; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Canagliflozin — One 300 mg over-encapsulated tablet taken orally (by mouth) once daily for 4 days during Part 1 and Part 2 (Sequence 1 [treatment period 2] or Sequence 2 [treatment period 1]).
  Other Names: Invokana
Drug: Dapagliflozin — One 10 mg over-encapsulated tablet taken orally once daily for 4 days during Part 2 (Sequence 1 [treatment period 1] or Sequence 2 [treatment period 2]).
  Other Names: Forxiga
  Arms: Part 2: Sequence 1 (Dapa/Cana); Part 2: Sequence 2 (Cana/Dapa)

SUMMARY:
The purpose of this study is to compare the pharmacodynamics (ie, how the drug affects the body) of canagliflozin with the pharmacodynamics of dapagliflozin.

DETAILED DESCRIPTION:
The study will be conducted as a 2-part study. Part 1 is an open-label pilot study (the investigator and the participants know the identity of the assigned treatment) in which 6 healthy volunteers will be given 300 mg of canagliflozin once daily for 4 consecutive days. The total study duration for each volunteer in Part 1 will be approximately 35 days (including a screening phase, an open-label treatment phase, and a follow-up phase). Part 2 will be a double-blind (neither the investigator nor volunteers know the identity of the assigned treatment), randomized (the treatment is assigned by chance), 2-period crossover study (all volunteers will receive each of the 2 treatments but in a different order) with a two-stage sequential group design.

Approximately 34 healthy volunteers will be participating in the first stage. After all the participants of the first stage will complete Part 2, and the results are analyzed, based on the first stage outcomes the study will be either terminated or will proceed to the second stage, which will be conducted using the same study method as in the first stage.

Potentially, up to 30 volunteers will participate in the second stage. A total number of participants in Part 2 will be up to 64.

Volunteers assigned to Treatment Sequence 1 will receive 10 mg of dapagliflozin once daily for 4 consecutive days (Period 1), and after a 12- to 14-day washout period (with no medication), 300 mg of canagliflozin once daily for 4 days (Period 2). Volunteers assigned to Treatment Sequence 2 will receive 300 mg of canagliflozin once daily for 4 days (Period 1), and after a 12- to 14-day washout period, 10 mg of dapagliflozin once daily for 4 consecutive days (Period 2). The total study duration for each volunteer in Part 2 will be up to approximately 65 days (including a screening phase, a baseline phase, a double-blind treatment phase, a washout period, and a follow-up phase).

Volunteers can participate in Part 1 or Part 2 of the study, but not in both parts. Canagliflozin and dapagliflozin are used for the treatment of type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have a body mass index (BMI = weight in kg/height in m2) between 20 and 27 kg/m2 (inclusive), and body weight >= 50 kg at Screening
* Volunteers must have a systolic blood pressure between 90 and 140 mmHg, inclusive, and a diastolic blood pressure no higher than 90 mmHg (based upon an average of 3 blood pressure readings at Screening)
* Volunteers must be non-smokers

Exclusion Criteria:

* Major surgery (eg, requiring general anesthesia) within 12 weeks before Screening, or planned during participation in the study, or within 2 weeks after the last dose of study drug administration, or volunteer will not have fully recovered from surgery during participation in the study; volunteers with planned surgical procedures to be conducted under local anesthesia may participate
* History of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening
* History of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at Screening
* History of, or currently active illness, considered to be clinically significant by the Investigator or any other illness that the Investigator considers should exclude the volunteer from the study or that could interfere with the interpretation of the study results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Between treatment difference in 24-hour mean renal threshold for glucose for canagliflozin (300 mg once daily for 4 days) compared to dapagliflozin (10 mg once daily for 4 days) | Day 4
  Renal threshold is defined as the plasma glucose concentration above which glucose is excreted in the urine.

SECONDARY OUTCOMES:
Percent change from baseline in postprandial glucose area under the curve at 0-2 hours post-dose on Day 4 following 300 mg of canagliflozin once daily for 4 days or 10 mg of dapagliflozin once daily for 4 days | Day -10 (Baseline) and Day 4
  Area under the concentration time curve (or area under the curve) is a measure of the body's exposure to glucose over a specific time period.
Number of volunteers with adverse events | Up to Day 65
  Adverse events will be used as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Neuss, Germany